CLINICAL TRIAL: NCT00358943
Title: Gaucher Disease Registry Protocol
Brief Title: International Collaborative Gaucher Group (ICGG) Gaucher Disease Registry & Pregnancy Sub-registry
Status: Recruiting | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DIREGC07009; ICGG Gaucher Registry (Other: Sanofi); U1111-1295-5844 (Registry Identifier: ICTRP)
Record Dates: First submitted 2006-07-12; First posted 2006-08-01 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Gaucher Disease; Cerebroside Lipidosis Syndrome; Glucocerebrosidase Deficiency Disease; Glucosylceramide Beta-Glucosidase Deficiency Disease
Keywords: Gaucher Disease; Glucocerebrosidase Deficiency Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients in ICGG Gaucher Registry: No experimental intervention is given. A patient with Gaucher Disease will undergo clinical assessments and receive standard of care treatment as determined by the patient's physician.
- Pregnant women with confirmed diagnosis of Gaucher disease: No experimental intervention is given. Pregnant women with confirmed diagnosis of Gaucher disease who are participating in the ICGG Gaucher Registry and consented to participate in the Gaucher Pregnancy Sub-registry, regardless of whether she is receiving disease-specific therapy and irrespective of the commercial product with which she may be treated.

SUMMARY:
The ICGG Gaucher Registry is an ongoing, international multi-center, strictly observational program that tracks the routine clinical outcomes for patients with Gaucher disease, irrespective of treatment status. No experimental intervention is involved; patients in the Registry undergo clinical assessments and receive care as determined by the patient's treating physician.

The objectives of the Registry are:

* To enhance understanding of the variability, progression, identification, and natural history of Gaucher disease, with the ultimate goal of better guiding and assessing therapeutic intervention.
* To assist the Gaucher medical community with the development of recommendations for monitoring patients, and to provide reports on patient outcomes, to optimize patient care.
* To characterize the Gaucher disease population.
* To evaluate the long-term effectiveness of imiglucerase and of eliglustat.

Gaucher Pregnancy Sub-registry: The primary objective of this Sub-registry is to track pregnancy outcomes, including complications and infant growth, in all women with Gaucher disease during pregnancy, regardless of whether they receive disease-specific therapy. No experimental intervention is given; thus a patient will undergo clinical assessments and receive standard of care treatment as determined by the patient's physician.If a patient consents to this Sub-registry, information about the patient's medical and obstetric history, pregnancy, and birth will be collected, and, if a patient consents to data collection for her infant, data on infant growth through month 36 postpartum will be collected.

ELIGIBILITY:
Inclusion Criteria:

ICGG Gaucher Registry

* All patients with a confirmed diagnosis of Gaucher disease are eligible for inclusion in the Registry. Confirmed diagnosis is defined as a documented β-glucocerebrosidase deficiency and/or mutation in the β-glucocerebrosidase gene.
* For all patients, appropriate patient authorization will be obtained.

Gaucher Pregnancy Sub-registry:

* be enrolled in the ICGG Gaucher Registry.
* be pregnant, or have been pregnant with appropriate medical documentation available.
* provide a signed informed consent and authorization form(s) to participate in the Sub-Registry prior to any Sub-Registry-related data collection being performed.

Exclusion Criteria:

- No exclusion criteria for participation in the ICGG Gaucher Registry and Sub-registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of Gaucher disease are eligible for inclusion in the ICGG Gaucher Registry.
  For Gaucher Pregnancy Sub-registry: It is recommended that pregnancy data be collected on all eligible women regardless of infant enrollment. In the event of patients having multiple pregnancies, data collection for each individual pregnancy is encouraged for all women enrolled in this Sub-registry.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 1991-04-01 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
ICGG Gaucher Registry: To provide the Gaucher medical community with recommendations for monitoring patients and to provide reports on patient outcomes to help optimize patient care | 42 years
Gaucher Pregnancy Sub-registry: To track pregnancy outcomes, including complications and infant growth, in all women with Gaucher disease during pregnancy, regardless of whether they receive disease-specific therapy, such as ERT with imiglucerase | 42 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Genzyme, a Sanofi Company
Locations (318):
- United States (85):
  - Phoenix Children's Hospital- Site Number : 840003, Phoenix, Arizona
  - University of Arizona- Site Number : 840015, Tucson, Arizona
  - Arkansas Childrens Hospital- Site Number : 840109, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences- Site Number : 840113, Little Rock, Arkansas
  - Tower Hematology/Oncology Medical Group- Site Number : 840056, Beverly Hills, California
  - University of California at Irvine- Site Number : 840036, Irvine, California
  - Southern California Permanente Medical Group- Site Number : 840108, Los Angeles, California
  - USC Health Sciences Center Dept of Genetics- Site Number : 840082, Los Angeles, California
  - Children's Hospital of Orange County- Site Number : 840074, Orange, California
  - Stanford Unviersity MC Dept of Genetics- Site Number : 840022, Palo Alto, California
  - UC Davis MIND Institute- Site Number : 840010, Sacramento, California
  - Kaiser Permanente Hospital- Site Number : 840042, Sacramento, California
  - University of California at San Diego- Site Number : 840007, San Diego, California
  - University of California at San Francisco- Site Number : 840051, San Francisco, California
  - Yale - Site Number : 840047, New Haven, Connecticut
  - Children's National Medical Center- Site Number : 840067, Washington D.C., District of Columbia
  - University Hematology Oncology- Site Number : 840075, Coral Springs, Florida
  - University of Florida Pediatrics Genetics- Site Number : 840121, Jacksonville, Florida
  - The Atwal Clinic- Site Number : 840112, Jacksonville, Florida
  - University Of Miami SOM- Site Number : 840006, Miami, Florida
  - University of Florida-Genetics- Site Number : 840096, Tampa, Florida
  - Pediatric Endocrine Associates- Site Number : 840017, Tampa, Florida
  - Emory University School of Medicine- Human Genetics- Site Number : 840060, Decatur, Georgia
  - University of Colorado at Denver Genetics- Site Number : 840068, Aurora, Illinois
  - Ann and Robert Lurie Children's Hospital- Site Number : 840011, Chicago, Illinois
  - Ann and Robert Lurie Children's Hospital- Site Number : 840013, Chicago, Illinois
  - Rush University Medical Center Genetics- Site Number : 840079, Chicago, Illinois
  - Indianapolis University School of Medicine- Site Number : 840027, Indianapolis, Indiana
  - University of Iowa- Site Number : 840032, Iowa City, Iowa
  - University of Louisville- Genetics- Site Number : 840030, Louisville, Kentucky
  - Tulane University Medical Center- Site Number : 840001, New Orleans, Louisiana
  - Maine Medical Center Pediatrics- Site Number : 840064, Portland, Maine
  - John Hopkins- Site Number : 840044, Baltimore, Maryland
  - Massachusetts General Hospital-Genetics- Site Number : 840062, Boston, Massachusetts
  - Boston Children's Hospital - PIN- Site Number : 840092, Boston, Massachusetts
  - University of Michigan Pediatrics- Site Number : 840107, Ann Arbor, Michigan
  - Children's Hospital of Michigan- Site Number : 840066, Detroit, Michigan
  - Spectrum for Health- Site Number : 840019, Grand Rapids, Michigan
  - Infusion Associates- Site Number : 840050, Grand Rapids, Michigan
  - Children's Health Care- Site Number : 840114, Minneapolis, Minnesota
  - Children's Hospital and Clinics of Minnesota- Site Number : 840046, Minneapolis, Minnesota
  - University of Minnesota Medical Center Pediatrics- Site Number : 840076, Minneapolis, Minnesota
  - University of Missouri Health System Department of Genetics- Site Number : 840031, Columbia, Missouri
  - Children's Mercy Hospital- Pediatrics- Site Number : 840063, Kansas City, Missouri
  - Washington University of St. Louis- Site Number : 840100, St Louis, Missouri
  - University of Nebraska Medical Center- Pediatrics- Site Number : 840084, Omaha, Nebraska
  - Children's Specialty Center of Nevada- Site Number : 840008, Las Vegas, Nevada
  - Cooper Health Center- Site Number : 840098, Camden, New Jersey
  - Joseph M. Sanzari Children's Hospital- Site Number : 840101, Hackensack, New Jersey
  - Atlantic Health System- Site Number : 840099, Morristown, New Jersey
  - St. Peter's University Hospital- Site Number : 840016, New Brunswick, New Jersey
  - St. Joseph's Children's Hospital- Site Number : 840057, Paterson, New Jersey
  - Northwell Health- Site Number : 840102, Manhasset, New York
  - New York University School Of Medicine- Site Number : 840040, New York, New York
  - Metropolitan Hospital Center- Site Number : 840110, New York, New York
  - Mt. Sinai School of Medicine- Site Number : 840005, New York, New York
  - Columbia University Irving Medical Center- Site Number : 840125, New York, New York
  - University of Rochester Medical Center SOM- Site Number : 840105, Rochester, New York
  - State University of New York- Site Number : 840052, Syracuse, New York
  - New York Medical College- Site Number : 840039, Valhalla, New York
  - Carolinas Medical Center Hospital- Site Number : 840065, Charlotte, North Carolina
  - Duke University Medical Center Genetics Dept- Site Number : 840037, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 840026, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 840119, Cleveland, Ohio
  - Cleveland Clinic Foundation Pediatrics- Site Number : 840048, Cleveland, Ohio
  - Nationwide Children's Hospital - PIN- Site Number : 840091, Columbus, Ohio
  - LSD Data Registry Site LLC- Site Number : 840094, Dublin, Ohio
  - Oregon Health & Science University (OHSU)- Site Number : 840080, Portland, Oregon
  - Penn State Health Milton South Hershey Medical Center- Site Number : 840126, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia HUP Medical Genetics- Site Number : 840089, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia- Site Number : 840034, Philadelphia, Pennsylvania
  - University of Pittsburgh- Site Number : 840023, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Genetics- Site Number : 840053, Providence, Rhode Island
  - Greenwood Genetcs- Site Number : 840055, Greenville, South Carolina
  - Vanderbilt University Hospital-Pediatrics- Site Number : 840049, Nashville, Tennessee
  - Baylor Research Center- Site Number : 840058, Dallas, Texas
  - Cook Children's Health Care System- Site Number : 840024, Fort Worth, Texas
  - University of Utah Department of Medical Genetics- Site Number : 840043, Salt Lake City, Utah
  - University of Virginia School of Medicine-Pediatrics- Site Number : 840078, Charlottesville, Virginia
  - O&O Alpan, LLC- Site Number : 840025, Fairfax, Virginia
  - Children's Hospital of the Kings Daughters- Site Number : 840072, Norfolk, Virginia
  - Seattle Children's Hospital- Site Number : 840028, Seattle, Washington
  - University Of Washington Medical Center- Site Number : 840059, Seattle, Washington
  - Multicare Health System ¿ Mary Bridge Childrens Hospital- Site Number : 840115, Tacoma, Washington
  - Children's Hospital of Wisconsin-Pediatrics- Site Number : 840054, Milwaukee, Wisconsin
- Argentina (7):
  - Investigational Site Number : 150661, CABA, Buenos Aires
  - Investigational Site Number : 032014, Ciudad de Buenos Aires, Buenos Aires
  - Investigational Site Number : 032003, La Plata, Buenos Aires
  - Investigational Site Number : 151085, Sarandí, Buenos Aires
  - Investigational Site Number : 032012, Buenos Aires
  - Investigational Site Number : 154176, Corrientes
  - Investigational Site Number : 032011, Córdoba
- Australia (9):
  - Investigational Site Number : 151431, Sydney, New South Wales
  - Investigational Site Number : 151069, Westmead, New South Wales
  - Investigational Site Number : 151010, Brisbane, Queensland
  - Investigational Site Number : 151491, Douglas, Queensland
  - Investigational Site Number : 151002, Adelaide, South Australia
  - Investigational Site Number : 151725, Hobart, Tasmania
  - Investigational Site Number : 151011, Clayton, Victoria
  - Investigational Site Number : 151008, Parkville, Victoria
  - Investigational Site Number : 151015, Murdoch, Western Australia
- Belgium (9):
  - Investigational Site Number : 150722, Antwerp
  - Investigational Site Number : 151156, Bruges
  - Investigational Site Number : 151796, Brussels
  - Investigational Site Number : 150944, Brussels
  - Investigational Site Number : 152345, Brussels
  - Investigational Site Number : 150517, Brussels
  - Investigational Site Number : 154285, Edegem
  - Investigational Site Number : 151134, Ghent
  - Investigational Site Number : 151668, Leuven
- Brazil (8):
  - Hospital das Clínicas da Universidade Federal do Paraná - HCUFPR- Site Number : 076010, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre- Site Number : 076007, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - PUC-Campinas- Site Number : 076012, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto- Site Number : 076001, Ribeirão Preto, São Paulo
  - Faculdade De Medicina - Unicamp- Site Number : 076005, Campinas
  - HEMORIO- Site Number : 076006, Rio de Janeiro
  - Instituto de Genética e Erros Inatos do Metabolismo- Site Number : 076002, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 076008, São Paulo
- Bulgaria (2):
  - Investigational Site Number : 100001, Sofia
  - Investigational Site Number : 151164, Sofia
- Canada (12):
  - Investigational Site Number : 124014, Calgary, Alberta
  - Investigational Site Number : 124002, Edmonton, Alberta
  - Investigational Site Number : 124010, Vancouver, British Columbia
  - Investigational Site Number : 124011, Vancouver, British Columbia
  - Investigational Site Number : 124019, Winnipeg, Manitoba
  - Investigational Site Number : 124022, Moncton, New Brunswick
  - Investigational Site Number : 124024, Kingston, Ontario
  - Investigational Site Number : 124005, Kingston, Ontario
  - Investigational Site Number : 124021, London, Ontario
  - Investigational Site Number : 124006, Toronto, Ontario
  - Investigational Site Number : 124013, Toronto, Ontario
  - Investigational Site Number : 124001, Sherbrooke, Quebec
- China (10):
  - Investigational Site Number : 151787, Beijing
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 156003, Beijing
  - Investigational Site Number : 152357, Guangzhou
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 152358, Hangzhou
  - Investigational Site Number : 152359, Hangzhou
  - Investigational Site Number : 157252, Nanjing
  - Investigational Site Number : 152356, Shanghai
  - Investigational Site Number : 150899, Shanghai
- Investigational Site Number : 170004, Bogotá, Colombia
- Croatia (3):
  - Investigational Site Number : 1910001, Zagreb
  - Investigational Site Number : 1910002, Zagreb
  - Investigational Site Number : 1910003, Zagreb
- Investigational Site Number : 150809, Prague, Czechia
- Investigational Site Number : 151229, København Ø, Denmark
- Investigational Site Number : 2140001, Santo Domingo, Dominican Republic
- Egypt (7):
  - Investigational Site Number : 818007, Al Mansurah
  - Investigational Site Number : 5748, Alexandria
  - Investigational Site Number : 9889, Ash Sharqiyah
  - Investigational Site Number : 9888, Asyut
  - Investigational Site Number : 9829, Cairo
  - Investigational Site Number : 8345, Cairo
  - Investigational Site Number : 9830, Cairo
- France (17):
  - Investigational Site Number : 250004, Besançon
  - Investigational Site Number : 250008, Bordeaux
  - Investigational Site Number : 250005, Brest
  - Investigational Site Number : 250014, Bron
  - Investigational Site Number : 250002, Caen
  - Investigational Site Number : 250001, Clichy
  - Investigational Site Number : 250003, Garches
  - Investigational Site Number : 250009, Lyon
  - Investigational Site Number : 250011, Marseille
  - Investigational Site Number : 2500013, Montpellier
  - Investigational Site Number : 250006, Nantes
  - Investigational Site Number : 250007, Paris
  - Investigational Site Number : 250010, Paris
  - Investigational Site Number : 250012, Rennes
  - Investigational Site Number : 250018, Strasbourg
  - Investigational Site Number : 250017, Toulouse
  - Investigational Site Number : 250016, Tours
- Germany (7):
  - Investigational Site Number : 151686, Berlin
  - Investigational Site Number : 150783, Düsseldorf
  - Investigational Site Number : 154150, Giessen
  - Investigational Site Number : 151369, Hamburg
  - Investigational Site Number : 151368, Hamburg
  - Investigational Site Number : 150031, Mainz
  - Investigational Site Number : 150432, Oberhausen
- Greece (4):
  - Investigational Site Number : 300002, Athens
  - Investigational Site Number : 300004, Athens
  - Investigational Site Number : 300003, Pátrai
  - Investigational Site Number : 300001, Thessaloniki
- Investigational Site Number : 344001, Kowloon, Hong Kong
- Hungary (4):
  - Investigational Site Number : 3480006, Budapest
  - Investigational Site Number : 3480003, Létavértes
  - Investigational Site Number : 3480007, Nyíregyháza
  - Investigational Site Number : 3480008, Székesfehérvár
- India (6):
  - Investigational Site Number : 356003, Ahmedabad
  - Investigational Site Number : 356004, Jaipur
  - Investigational Site Number : 356001, Kolkata
  - Investigational Site Number : 356005, Mumbai
  - Investigational Site Number : 3560006, Secunderabad
  - Investigational Site Number : 356002, Vellore
- Investigational Site Number : 360001, Jakarta, Indonesia
- Israel (3):
  - Investigational Site Number : 3760003, Haifa
  - Investigational Site Number : 3760001, Jerusalem
  - Investigational Site Number : 3760002, Petah Tikva
- Italy (12):
  - Investigational Site Number : 380007, Rome, Roma
  - Investigational Site Number : 380014, Sassari, Sardinia
  - Investigational Site Number : 380008, Catania
  - Investigational Site Number : 380009, Florence
  - Investigational Site Number : 380006, Genova
  - Investigational Site Number : 380004, Milan
  - Investigational Site Number : 380005, Modena
  - Investigational Site Number : 380002, Monza
  - Investigational Site Number : 380011, Monza
  - Investigational Site Number : 380010, Napoli
  - Investigational Site Number : 380003, Padua
  - Investigational Site Number : 380001, Udine
- Japan (4):
  - Investigational Site Number : 153205, Abeno-ku, Osaka
  - Investigational Site Number : 153203, Yonago-shi, Tottori
  - Investigational Site Number : 153217, Chiba
  - Investigational Site Number : 153204, Tokyo
- Investigational Site Number : 4000001, Amman, Jordan
- Investigational Site Number : 154225, Kuwait City, Kuwait
- Lebanon (2):
  - Investigational Site Number : 422001, Beirut
  - Investigational Site Number : 4220004, Beirut
- Investigational Site Number : 154237, Vilnius, Lithuania
- Malaysia (2):
  - Investigational Site Number : 458002, Kuala Lumpur
  - Investigational Site Number : 458001, Kuala Pahang
- Netherlands (2):
  - Investigational Site Number : 150149, Amsterdam
  - Investigational Site Number : 151171, Amsterdam
- Pakistan (2):
  - Investigational Site Number : 154264, Karachi
  - Investigational Site Number : 154266, Lahore
- Peru (2):
  - Investigational Site Number : 604001, Arequipa
  - Investigational Site Number : 604002, Callao
- Investigational Site Number : 608001, Manila, Philippines
- Investigational Site Number : 150575, Warsaw, Poland
- Portugal (3):
  - Investigational Site Number : 620003, Coimbra
  - Investigational Site Number : 620004, Lisbon
  - Investigational Site Number : 620009, Ponta Delgada
- Romania (3):
  - Investigational Site Number : 642001, Cluj-Napoca
  - Investigational Site Number : 151188, Cluj-Napoca
  - Investigational Site Number : 642002, Cluj-Napoca
- Russia (2):
  - Investigational Site Number : 643001, Moscow
  - Investigational Site Number : 643002, Saint Petersburg
- Saudi Arabia (3):
  - Investigational Site Number : 682002, Al Mubarraz
  - Investigational Site Number : 682003, Jeddah
  - Investigational Site Number : 682004, Mecca
- Serbia (5):
  - Investigational Site Number : 688001, Belgrade
  - Investigational Site Number : 688002, Belgrade
  - Investigational Site Number : 688003, Belgrade
  - Investigational Site Number : 688005, Belgrade
  - Investigational Site Number : 688004, Niš
- Investigational Site Number : 702001, Singapore, Singapore
- Investigational Site Number : 703001, Bratislava, Slovakia
- South Africa (3):
  - Investigational Site Number : 154138, Johannesburg
  - Investigational Site Number : 710-003, Johannesburg
  - Investigational Site Number : 150346, Sandton
- South Korea (7):
  - Investigational Site Number : 154208, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 153180, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153196, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153191, Daejeon
  - Investigational Site Number : 151149, Seoul
  - Investigational Site Number : 153212, Seoul
  - Investigational Site Number : 153222, Seoul
- Spain (17):
  - Investigational Site Number : 154146, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 153237, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 154147, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 154119, Alcorcón, Madrid
  - Investigational Site Number : 153213, Vigo, Pontevedra [Pontevedra]
  - Investigational Site Number : 153215, Seville, Sevilla
  - Investigational Site Number : 153219, Seville, Sevilla
  - Investigational Site Number : 154163, Madrid
  - Investigational Site Number : 154236, Madrid
  - Investigational Site Number : 151524, Madrid
  - Investigational Site Number : 153251, Madrid
  - Investigational Site Number : 154199, Madrid
  - Investigational Site Number : 154160, Madrid
  - Investigational Site Number : 154145, Sabadell
  - Investigational Site Number : 154205, Valencia
  - Investigational Site Number : 154238, Zaragoza
  - Investigational Site Number : 153216, Zaragoza
- Sweden (3):
  - Investigational Site Number : 154095, Borås
  - Investigational Site Number : 151726, Malmo
  - Investigational Site Number : 154092, Norrköping
- Switzerland (4):
  - Investigational Site Number : 157237, Aarau
  - Investigational Site Number : 157045, Bern
  - Investigational Site Number : 157244, Lausanne
  - Investigational Site Number : 157241, Zurich
- Taiwan (14):
  - Investigational Site Number : 151500, Chiayi City
  - Investigational Site Number : 154093, Chiayi City
  - Investigational Site Number : 152152, Hualien City
  - Investigational Site Number : 152244, Kaohsiung City
  - Investigational Site Number : 152246, Kaohsiung City
  - Investigational Site Number : 151534, New Taipei City
  - Investigational Site Number : 151181, Taichung
  - Investigational Site Number : 151179, Taichung
  - Investigational Site Number : 153248, Tainan
  - Investigational Site Number : 152153, Tainan
  - Investigational Site Number : 151182, Taipei
  - Investigational Site Number : 152321, Taipei
  - Investigational Site Number : 152226, Taipei
  - Investigational Site Number : 153158, Tao Yuan County
- Thailand (4):
  - Investigational Site Number : 764003, Bangkok
  - Investigational Site Number : 764004, Bangkok
  - Investigational Site Number : 764001, Bangkok
  - Investigational Site Number : 764005, Khon Kaen
- Turkey (Türkiye) (7):
  - Investigational Site Number : 792006, Adana
  - Investigational Site Number : 792005, Ankara
  - Investigational Site Number : 792001, Ankara
  - Investigational Site Number : 792002, Ankara
  - Investigational Site Number : 792004, Istanbul
  - Investigational Site Number : 792007, Izmir
  - Investigational Site Number : 792003, Malatya
- Investigational Site Number : 7840001, Dubai, United Arab Emirates
- United Kingdom (8):
  - Investigational Site Number : 151340, Cambridge, Cambridgeshire
  - Investigational Site Number : 152287, Birmingham, England
  - Investigational Site Number : 152361, Salford, Manchester
  - Investigational Site Number : 154240, Birmingham
  - Investigational Site Number : 151123, London
  - Investigational Site Number : 151646, London
  - Investigational Site Number : 150303, London
  - Investigational Site Number : 150455, Manchester
- Vietnam (2):
  - Investigational Site Number : 154212, Hanoi
  - Investigational Site Number : 704002, Ho Chi Minh City

REFERENCES:
- [Background] El-Beshlawy A, Tylki-Szymanska A, Vellodi A, Belmatoug N, Grabowski GA, Kolodny EH, Batista JL, Cox GF, Mistry PK. Long-term hematological, visceral, and growth outcomes in children with Gaucher disease type 3 treated with imiglucerase in the International Collaborative Gaucher Group Gaucher Registry. Mol Genet Metab. 2017 Jan-Feb;120(1-2):47-56. doi: 10.1016/j.ymgme.2016.12.001. Epub 2016 Dec 6. PMID 28040394
- [Background] Mistry PK, Batista JL, Andersson HC, Balwani M, Burrow TA, Charrow J, Kaplan P, Khan A, Kishnani PS, Kolodny EH, Rosenbloom B, Scott CR, Weinreb N. Transformation in pretreatment manifestations of Gaucher disease type 1 during two decades of alglucerase/imiglucerase enzyme replacement therapy in the International Collaborative Gaucher Group (ICGG) Gaucher Registry. Am J Hematol. 2017 Sep;92(9):929-939. doi: 10.1002/ajh.24801. Epub 2017 Jul 7. PMID 28569047
- [Background] Weinreb NJ, Goldblatt J, Villalobos J, Charrow J, Cole JA, Kerstenetzky M, vom Dahl S, Hollak C. Long-term clinical outcomes in type 1 Gaucher disease following 10 years of imiglucerase treatment. J Inherit Metab Dis. 2013 May;36(3):543-53. doi: 10.1007/s10545-012-9528-4. Epub 2012 Sep 14. PMID 22976765
- [Derived] Ain NU, Vaishnaw M, Mistry PK. Natural-History Mapping of Lysosomal Storage Disorders (LSDs): Gaucher Disease as a Model for Precision Care. J Inherit Metab Dis. 2026 Jan;49(1):e70128. doi: 10.1002/jimd.70128. PMID 41527340
- [Derived] Rosenbloom BE, Cappellini MD, Weinreb NJ, Dragosky M, Revel-Vilk S, Batista JL, Sekulic D, Mistry PK. Cancer risk and gammopathies in 2123 adults with Gaucher disease type 1 in the International Gaucher Group Gaucher Registry. Am J Hematol. 2022 Oct;97(10):1337-1347. doi: 10.1002/ajh.26675. Epub 2022 Aug 24. PMID 36054609
- [Derived] Weinreb NJ, Camelo JS Jr, Charrow J, McClain MR, Mistry P, Belmatoug N; International Collaborative Gaucher Group (ICGG) Gaucher Registry (NCT00358943) investigators. Gaucher disease type 1 patients from the ICGG Gaucher Registry sustain initial clinical improvements during twenty years of imiglucerase treatment. Mol Genet Metab. 2021 Feb;132(2):100-111. doi: 10.1016/j.ymgme.2020.12.295. Epub 2021 Jan 8. PMID 33485799
- [Derived] Weinreb NJ, Kaplan P. The history and accomplishments of the ICGG Gaucher registry. Am J Hematol. 2015 Jul;90 Suppl 1:S2-5. doi: 10.1002/ajh.24054. No abstract available. PMID 26096743
- [Derived] Buyers RP, Collin-Histed T. Foreword. Am J Hematol. 2015 Jul;90 Suppl 1:S1. doi: 10.1002/ajh.24053. No abstract available. PMID 26096740